CLINICAL TRIAL: NCT04075955
Title: FORESIGHT: Feasibility of Olanzapine at REduced doSe in hIGHly Emetogenic chemoTherapy: a Randomised Controlled Trial Against Aprepitant in Triple Therapy
Brief Title: Feasibility of Olanzapine at REduced doSe in hIGHly Emetogenic chemoTherapy
Acronym: FORESIGHT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CR-CSSS Champlain-Charles-Le Moyne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-389
Record Dates: First submitted 2019-05-10; First posted 2019-09-03 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Chemotherapy-induced Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Olanzapine; Aprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study treatment group (Experimental): Olanzapine in combination with ondansetron and dexamethasone
  Interventions: Drug: Zyprexa® (OLANZapine 5MG)
- Standard treatment group (Active Comparator): Aprepitant in combination with ondansetron and dexamethasone
  Interventions: Drug: Emend® (Aprepitant)

INTERVENTIONS:
Drug: Zyprexa® (OLANZapine 5MG) — Olanzapine 5mg orally at bedtime for 4 days (starting the day before the chemotherapy)
  Ondansetron 16mg orally pre-chemotherapy on day 1
  Dexamethasone 12mg orally pre-chemotherapy on day 1
  Dexamethasone 8mg orally twice a day for 6 doses (starting on the morning of day 2)
  Other Names: Zyprexa®
  Arms: Study treatment group
Drug: Emend® (Aprepitant) — Aprepitant 125mg orally pre-chemotherapy on day 1, then 80mg orally once daily on days 2 and 3
  Ondansetron 16mg orally pre-chemotherapy on day 1
  Dexamethasone 12mg orally pre-chemotherapy on day 1
  Dexamethasone 8mg orally once daily for 3 doses (starting on the morning of day 2)
  Other Names: Emend®
  Arms: Standard treatment group

SUMMARY:
Olanzapine is frequently used off-label as an adjunct antiemetic in clinical oncology settings. North American oncology guidelines recommend it as salvage therapy and as add-on to the standard triple regimen; some suggest it may also be effective as an initial triple therapy (olanzapine replacing the NK-1 antagonist) based on phase II and III trials.

This prospective, multi-center, open-label study aims to evaluate the feasibility of a large scale randomised controlled trial to compare the effectiveness and tolerability of 5mg orally once daily olanzapine in triple antiemetic therapy versus the standard treatment of aprepitant + ondansetron + dexamethasone in treatment-naive patients receiving the first cycle of a highly emetogenic chemotherapy. Secondary outcomes include effectiveness, tolerability and quality of life assessments. Effectiveness will be measured with complete response and complete remission rates in each treatment arms. Tolerability and patient quality of life will be evaluated with a standardised side effect form and validated questionnaires; ESAS-R and FLIE.

The role of olanzapine-based triple therapy in prevention of chemotherapy-induced nausea and vomiting remains founded on low-quality evidence. To the investigator's knowledge, this study will be the first large scale direct comparison of 5mg olanzapine versus aprepitant in triple therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving a first cycle of highly emetogenic chemotherapy (or having received one more than 2 years prior to randomisation) at the oncology outpatient clinic at Charles LeMoyne or Haut-Richelieu hospital between April 29th and September 20th 2019.
* 18 years old and over
* Patient receiving highly emetogenic chemotherapy
* ECOG from 0 to 2 inclusively
* Creatinine clearance ≥ 30ml/min; total bilirubin ≤ 1.5 x ULN, AST/ALT ≤ 3.0 x ULN
* Patient without electrolytic imbalance or corrected imbalance
* Signed written and informed consent

Exclusion Criteria:

* Patient doesn't speak french or english
* Patient to receive treatment whose protocol includes a second dose of highly emetogenic chemotherapy before day 6 of the cycle
* Patient to receive chemotherapy treatment that already contains corticosteroids (dexamethasone or prednisone) given as antineoplastic
* Nausea or vomiting present ≤ 24h before randomisation
* Untreated brain metastases
* Severe cognitive disorder or dementia or inability to properly understand or document the presence of nausea or vomiting or the use of salvage therapy
* History of uncontrolled cardiac arrhythmia, unstable angina or known QT prolongation (> 500ms)
* Uncontrolled diabetes
* Patient to receive abdominal radiotherapy during the first cycle of chemotherapy
* Bowel obstruction, intestinal ileus or ascites present at cycle 1
* Chronic alcoholism
* Severe uncontrolled psychologic disorder
* Patient taking antipsychotic treatment on a regular basis
* Patient taking drugs with a contraindication when administered concurrently with one of the protocol drugs
* Dysphagia (incapacity to swallow the pills included in the study)
* Hypersensitivity, severe reaction or allergy to one of the study treatments
* Participation in another research protocol
* Pregnancy or breastfeeding
* Subject that does not have a valid phone ou email address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients recruited | 5 months
  At least 60 patients over 5 months meet the eligibility criteria and agree to participate.
Eligible patients' interest to participate | 5 months
  At least 35% of all eligible patients agree to participate
Completion of the diary | 5 months
  At least 75% of recruited patients complete 100% of their patient diary.
Cost | 5 months
  The total cost of the study does not exceed 10,000$
Number of centres | 5 months
  The study can be done at two sites.

SECONDARY OUTCOMES:
Compare effectiveness of olanzapine 5mg versus standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy in regard of proportion of participant with complete response in the overall phase. | 0 to 120 hours
  Overall phase was defined as 0 to 120 hours following initiation of chemotherapy.
  Complete response was defined as no nausea, no vomiting and no rescue therapy. Intensity of nausea episodes will be measured with a 0 to 10 visual scale. Intensity of vomiting episodes will be measured with a 0 to 10 visual scale.
Compare effectiveness of olanzapine 5mg versus standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy in regard of proportion of participant with complete remission in the overall phase. | 0 to 120 hours
  Overall phase was defined as 0 to 120 hours following initiation of chemotherapy.
  Complete remission was defined as no vomiting and no rescue therapy. Intensity of vomiting episodes will be measured with a 0 to 10 visual scale.
Compare tolerability of olanzapine 5mg versus standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy in regard of prevalence of adverse events due to the antiemetic therapy in each arm. | During the complete duration of the first cycle of chemotherapy (1 cycle is 14 to 28 days)
  Proportion of patients who experienced adverse events associated with each of the treatment arms. Adverse events obtained according to the ESAS-R questionnaire and a follow-up interview at the second cycle of chemotherapy.
  Definition and gradation of adverse events would be following the Common Terminology Criteria for Adverse Events (CTCAE) 5th edition.
Compare patient's assessment of quality of life between those receiving olanzapine 5mg and those receiving standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy. | 0 to 120 hours
  Quality of life score obtained according to the FLIE questionnaire

OTHER OUTCOMES:
Compare effectiveness of olanzapine 5mg versus standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy in regard of proportion of participant with complete response in the acute phase. | 0 to 24 hours
  Acute phase was defined as 0 to 24 hours following initiation of chemotherapy. Complete response was defined as no nausea, no vomiting and no rescue therapy. Intensity of nausea episodes will be measured with a 0 to 10 visual scale. Intensity of vomiting episodes will be measured with a 0 to 10 visual scale.
Compare effectiveness of olanzapine 5mg versus standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy in regard of proportion of participant with complete response in the delayed phase. | 24 to 120 hours
  Delayed phase was defined as 24 to 120 hours following initiation of chemotherapy.
  Complete response was defined as no nausea, no vomiting and no rescue therapy. Intensity of nausea episodes will be measured with a 0 to 10 visual scale. Intensity of vomiting episodes will be measured with a 0 to 10 visual scale.
Compare effectiveness of olanzapine 5mg versus standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy in regard of proportion of participant with complete remission in the acute phase. | 0 to 24 hours
  Acute phase was defined as 0 to 24 hours following initiation of chemotherapy. Complete remission was defined as no vomiting and no rescue therapy. Intensity of vomiting episodes will be measured with a 0 to 10 visual scale.
Compare effectiveness of olanzapine 5mg versus standard aprepitant in a triple antiemetic therapy in patients receiving a first cycle of highly emetogenic chemotherapy in regard of proportion of participant with complete remission in the delayed phase. | 24 to 120 hours
  Delayed phase was defined as 24 to 120 hours following initiation of chemotherapy.
  Complete remission was defined as no vomiting and no rescue therapy. Intensity of vomiting episodes will be measured with a 0 to 10 visual scale.
Compare rate of continuation of the same antiemetic regimen at cycle 2 between those receiving olanzapine 5mg and those receiving standard aprepitant in a triple antiemetic therapy. | 14 to 28 days
  Proportion of patients who desire to continue the same regimen at the end of the first cycle of chemotherapy (each cycle is usually between 14 to 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Prady, Md, Principal Investigator — CR-CISSS
Locations (1):
- Hôpital Charles-LeMoyne, Greenfield Park, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Prévention et traitement des nausées et vomissements induits par la chimiothérapie ou la radiothérapie chez l'adulte (Guide du CEPO) — http://www.msss.gouv.qc.ca/inc/documents/ministere/lutte-contre-le-cancer/guides-cepo-pdf/CEPO-Anti%C3%A9m%C3%A9tiques_MAJ_(2012-11-08).pdf
- See also: Olanzapine for the Prevention of Chemotherapy-Induced Nausea and Vomiting in Patients Receiving Highly or Moderately Emetogenic Chemotherapy: A Randomized, Double-Blind, Placebo-Controlled Study by Mizukami (2014) — http://www.ncbi.nlm.nih.gov/pubmed/23856100
- See also: Olanzapine for the prevention and treatment of cancer-related nausea and vomiting in adults. (Cochrane review 2018) — https://pubmed.ncbi.nlm.nih.gov/30246876/
- See also: Olanzapine Versus Aprepitant for the Prevention of Chemotherapy-Induced Nausea and Vomiting: A Randomized Phase III Trial by Navari (2011) — http://www.ncbi.nlm.nih.gov/pubmed/22024310
- See also: Olanzapine-Based Triple Regimens Versus Neurokinin-1 Receptor Antagonist-Based Triple Regimens in Preventing Chemotherapy-Induced Nausea and Vomiting Associated with Highly Emetogenic Chemotherapy: A Network Meta-Analysis (Zhang 2018) — http://www.ncbi.nlm.nih.gov/pubmed/29330211
- See also: Olanzapine for chemotherapy-induced nausea and vomiting: systematic review and meta-analysis (Chelkeba 2017) — http://www.ncbi.nlm.nih.gov/pubmed/28503222
- See also: Efficacy of olanzapine for the prophylaxis of chemotherapy-induced nausea and vomiting: a meta-analysis (Yang 2017) — http://www.ncbi.nlm.nih.gov/pubmed/28112422
- See also: A meta-analysis of olanzapine for the prevention of chemotherapy-induced nausea and vomiting (Wang 2014) — http://ncbi.nlm.nih.gov/pubmed/24770591
- See also: A double-blind randomized phase II dose-finding study of olanzapine 10 mg or 5 mg for the prophylaxis of emesis induced by highly emetogenic cisplatin-based chemotherapy by Yanai (2018) — http://www.ncbi.nlm.nih.gov/pubmed/29039073
- See also: Antiemetics: American Society of Clinical Oncology Clinical Practice Guideline Update 2017 — http://ascopubs.org/doi/abs/10.1200/JCO.2017.74.4789
- See also: Functional Living Index - Emesis (FLIE questionnaire) — https://eprovide.mapi-trust.org/instruments/functional-living-index-emesis
- See also: A tutorial on pilot studies: the what, why and how — http://bmcmedresmethodol.biomedcentral.com/articles/10.1186/1471-2288-10-1
- See also: Clinical research of Olanzapine for prevention of chemotherapy-induced nausea and vomiting — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC2761865/
- See also: Efficacy of olanzapine for the prophylaxis and rescue of chemotherapy-induced nausea and vomiting (CINV): a systematic review and meta-analysis (Chiu 2016) — http://ncbi.nlm.nih.gov/pubmed/26768437